CLINICAL TRIAL: NCT05204173
Title: Efficacy and Safety of Sintilimab Combined Intraperitoneal and Intravenous Paclitaxel Plus Oral S-1 in Gastric Cancer Patients With Peritoneal Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, zhuzhenggang, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRAGON-09
Record Dates: First submitted 2021-12-25; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Gastric Cancer Stage IV; Peritoneal Metastases
Keywords: Gastric cancer; Peritoneal metastasis; Paclitaxel; Sintilimab; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal (Experimental): Sintilimab 200mg intravenous (IV) infusion on day 1, PTX 50 mg/m2 IV and PTX 20 mg/m2 intraperitoneal infusion on Days 1 and 8 plus oral S-1 80 mg/m2 for 14 consecutive days every 3 weeks.
  Interventions: Drug: sintilimab, paclitaxel and S-1

INTERVENTIONS:
Drug: sintilimab, paclitaxel and S-1 — Sintilimab 200mg intravenous (IV) infusion on day 1, PTX 50 mg/m2 IV and PTX 20 mg/m2 intraperitoneal infusion on Days 1 and 8 plus oral S-1 80 mg/m2 for 14 consecutive days with one week rest.

SUMMARY:
In this phase 2 study, we combined sintilimab, paclitaxel and S-1 as regimen to treat gastric cancer patients with peritoneal metastasis. We are aim to estimate the efficacy and safety of this regimen in the phase 2 study.

DETAILED DESCRIPTION:
Gastric cancer patients enrolled in this a phase 2 study received sintilimab (200mg intravenously on day 1), paclitaxel (PTX) (20 mg/m2 intraperitoneally and 50 mg/m2 intravenously on days 1 and 8) plus oral S-1 (80 mg/m2 for 14 consecutive days) every 3 weeks. The primary endpoint is 1-year survival rate. Secondary endpoints are adverse events, R0 resection rate, 3-year overall survival (OS), and 3-year progressive free survival. Adverse events are monitored and graded according to the Common Terminology Criteria for Adverse Events version 4.0.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric adenocarcinoma;
2. Peritoneal metastases from gastric cancer requiring definitive diagnosis by laparoscopy, and without gastric outflow tract obstruction and intestinal obstruction;
3. Written (signed) informed consent;
4. Age ≥ 18 years at registration;
5. Eastern Cooperative Oncology Group (ECOG) score ≤ 2;
6. Expected life expectancy > 3 months;
7. Adequate bone marrow, liver, and renal functions. absolute neutrophil count of ≥1.5×109/L; absolute neutrophil count of ≥1.5×109/L; platelet count of ≥100×109/L; hemoglobin ≥90g/L; bilirubin of <1.5×upper limit of normal [ULN]; alanine aminotransferase and aspartate aminotransferase of <2.5×ULN; serum creatinine of ≤1.5×ULN; creatinine clearance of >50 mL/min; TSH ≤1×ULN (if abnormal, T3 and T4 levels should be inspected at the same time, if T3 and T4 levels are normal, they can be included in the group); APTT ≤1.5×ULN and INR ≤1.5×ULN; myocardial enzymogram ≤1×ULN.

Exclusion Criteria:

1. Confirmed of evidence of distant metastasis other than peritoneal metastasis (e.g.liver metastasis, lung metastasis, para-aortic lymph node metastasis, etc.);
2. During pregnancy, within 28 days of post parturition, or during lactation;
3. Synchronous or metachronous (within 5 years) malignancies.
4. Severe mental disease, uncontrolled epilepsy, or central nervous system disease;
5. Clinically severe (i.e. active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or arrhythmia requiring drug intervention, or a history of myocardial infarction in the last 12 months;
6. Upper gastrointestinal obstruction or abnormal physiological function or malabsorption syndrome may affect S-1 absorbers;
7. Known peripheral neuropathy (> NCI-CTC AE 1). However, patients with only disappearance of deep tendon reflex (DTR) need not be excluded;
8. Patients on steroid or immunosuppressant treatment after organ transplant;
9. Patients with severe uncontrolled recurrent infections or other severe uncontrolled concomitant disease;
10. Moderate or severe renal damage [creatinine clearance ≤ 50 ml/min], or serum creatinine > upper limit of normal (ULN), 115 μmol/L;
11. Known dihydropyrimidine dehydrogenase (DPD) deficiency;
12. Anaphylaxis to paclitaxel or any research drug ingredient.
13. Active autoimmune disease or history of refractory autoimmune disease; Subjects with hypothyroidism requiring only hormone replacement therapy and skin diseases without systemic treatment (such as vitiligo, psoriasis or alopecia) can be selected;
14. HIV antibody positive, active hepatitis B or C (hepatitis B: HBsAg positive and HBV DNA ≥10 copies/ml; hepatitis C: HCV antibody and HCV-RNA positive, requiring antiviral treatment at the same time);
15. Steroid or other systemic immunosuppressive therapy was used 14 days before admission, excluding local or physiological doses of systemic glucocorticoids (eg. no more than 10mg/day of prednisone or other glucocorticoids of equivalent dose) by nasal spray, inhalation or other routes, or hormones used to prevent allergy of contrast agents;
16. Uncontrolled arrhythmia and myocardial infarction within 12 months before admission or active tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
1-year survival rate | 12 months

SECONDARY OUTCOMES:
Number of participants experiencing clinical and laboratory adverse events (AEs) | 24 months
R0 resection rate | 24 months
3-year overall survival (OS) | 36 months
3-year progressive free survival (PFS) | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Yuan H, Lu S, Sun DB, Yao XX, Liu WT, Zheng YN, Hua ZC, Ni ZT, He CY, Wang ZQ, Zhang J, Liu D, Jiang C, Li C, Zhang J, Yan M, Yang ZY, Shi M, Zhu ZG, Yan C. Intraperitoneal and intravenous paclitaxel plus S-1 and sintilimab as first-line treatment for gastric cancer with peritoneal metastasis: a single-arm phase 2 trial (DRAGON-09). EClinicalMedicine. 2025 Dec 29;91:103731. doi: 10.1016/j.eclinm.2025.103731. eCollection 2026 Jan. PMID 41542221
- [Derived] Yuan H, Lu S, Shi M, Yang Z, Liu W, Ni Z, Yao X, Hua Z, Feng R, Zheng Y, Wang Z, Sah BK, Chen M, Zhu Z, He C, Li C, Zhang J, Yan C, Yan M, Zhu Z. Sintilimab combined neoadjuvant intraperitoneal and systemic chemotherapy in gastric cancer with peritoneal metastasis. Future Oncol. 2023 Dec;19(38):2517-2523. doi: 10.2217/fon-2022-0738. Epub 2023 May 22. PMID 37212686